CLINICAL TRIAL: NCT02345655
Title: Impact of On-site Evaluation of Substances Consumption on Opiate Maintenance in the Context of Family Practice
Brief Title: On-site Evaluation of Substances Consumption on Opiate Maintenance
Acronym: ESUB-MG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/13/7049; 2014-A00393-44 (Other: ID-RCB)
Record Dates: First submitted 2014-05-14; First posted 2015-01-26 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Opiate Addiction
Keywords: Substances consumption; Opiate; Family practice
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urine Drug Testing (Experimental): GPs of the intervention group will dedicate an average 5 minutes during the consult to perform OS-UDT. Patients will be asked to collect a urine sample at the GP's medical office. GP will read and communicate the results immediately to the patients. GPs will keep free of their management according to OS-UDT results.
  Interventions: Procedure: urine drug testing
- No test (Other): Patients will not have to performed the OS-UDT test
  Interventions: Other: no test

INTERVENTIONS:
Procedure: urine drug testing — Performed a OS-UDT test in general practice on patients starting buprenorphine
  Arms: Urine Drug Testing
Other: no test — normal procedure decided by the general practitioner
  Arms: No test

SUMMARY:
In France, General Practitioners (GPs) are widely involved in opiate maintenance treatment (OMT) by initially prescribing buprenorphine and monitoring patients under buprenorphine and methadone. Number of treated patients is around 150,000 with 75% of them treated by buprenorphine. Among the guidelines for improving OMT, urine testing is mandatory for initiating methadone, whereas it is recommended for initiating buprenorphine and during follow-up. Urine drug tests are based on immunoassay techniques and enable a qualitative analysis of the recent drug consumption, with detection based on designated thresholds, allow a better appraisal of drug exposure, before initiating and during OMT. While intrinsic diagnostic value of these tests is already demonstrated, the consequences of carrying out these tests on OMT have not been clearly established. Some studies suggest that patients exposed to drug tests may have a better OMT retention and in patients treated by methadone, performing urine screening tests has been shown to be associated with a mortality risk reduction in a Scottish retrospective cohort of opioid addicts. Actually, despite the recommendations to perform these tests, few GP prescribe tests, and few patients are regularly screened. Availability of commercial kits for urine drug testing in the medical office should improve their utilisation.

The widespread of urine drug screening tests use in ambulatory care is a reality for some GPs working in addictology networks. Despite a global benefit reported in the literature with a better control in prescribing OMT and a better patients' adherence, as far as the investigators know, no study has yet explored the impact of the use of urine drug screening test in decision making in general practice with an intervention study.

DETAILED DESCRIPTION:
In a retrospective cohort study of methadone users performed through data obtained from a primary care prescription registry in Tayside, Scotland, McCowan et al examined the interaction of patient related factors and prescribing factors at the individual level and assess their independent impact on the risk of both all-cause mortality and drug dependent cause specific mortality (McCowan, Kidd et al. 2009). Overall, 181 (8%) people died among 2378 subjects with a median follow-up of 4.38 years. Overuse of methadone, history of psychiatric admission, and increasing comorbidity were all associated with an increase in all-cause mortality. Longer duration of use (adjusted hazard ratio 0.95, 0.94 to 0.96), history of having urine tested (0.33, 0.22 to 0.49), and increasing time since last filled prescription were protective in relation to all-cause mortality. These factors are likely to be markers of people who are stabilised on maintenance treatment and engaged in monitoring procedures or who have successfully completed a methadone treatment reduction programme. This community based study gives a clear indication of the prescribing, monitoring, and management of patients in OMT and the subsequent impact on all cause and drug dependent mortality. This study provides evidence that recommendations on best practice (including specifically performing UDS) improve patients' outcomes.

Using data from the French "Methaville" trial, Roux et al (Roux, Michel et al. 2012; Roux, Lions et al. 2013) investigated the effect of pre-treatment and in-treatment factors on long-term non-adherence to this OMT. Four pre-treatment predictors of non-adherence were identified: being female, not having stable housing, alcohol consumption and cocaine use. These findings highlight the need to appropriately assess psychoactive drug use when starting OMT, and urine drug testing should be consider as a way to reach this aim.

On the basis of the literature, one would suppose that carrying out UDS would provide an improvement in the management of patients with abuse or addiction and would be helpful, particularly in community office-based settings, as office-based management of opioid dependence grows up (Walley, Alperen et al. 2008). Despite the lack of significant evidence of efficacy, UDS are recommended to assess the use of psychoactive substances when abuse or addiction is suspected.

ELIGIBILITY:
INCLUSION CRITERIA

* For GPs:Professional criteria: to practice as a GP, to be in activity, to practice in general ambulatory practice (in a medical office), to regularly manage patients treated with buprenorphine, to be registered in sector 1, consent for participating to the study
* For patients:

Aged 18 years-old or more, to consult for starting buprenorphine or OMT:

* any patient previously treated by buprenorphine or buprenorphine-naloxone but with his/her treatment interrupted for at least 2 months will be considered as a candidate for a new treatment with buprenorphine or buprenorphine-naloxone
* any patient previously exposed to opiate maintenance drug obtained illegally "in the street" will not be as treated affiliated to a health insurance scheme, not opposed to participate

EXCLUSION CRITERIA

- For patients: to consult for continuing buprenorphine or for another complain related, to opiate substitution treatment, to be known and yet managed by the GP for an opiate substitutive treatment, to have started buprenorphine in a specialized centre or in a hospital, to be treated with methadone, to be treated with methadone and asking a switch toward buprenorphine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Impact of on-site urine drug screening tests | 6 months
  The main objective will be to assess the impact of on-site urine drug screening tests in general practice compared to routine medical care on OMT retention at six months in opioid-dependent patients initiating buprenorphine.

SECONDARY OUTCOMES:
Acceptability of OS-UDT (One-site Urine Drug Testing) by patients and GPs | 6 months
  To assess if patients and GPs accept to performed the One-Site Urine Drug Testing
Patient's adherence to buprenorphine (duration and dose) | 6 months
  General Practitioner will assessed if patients follow their treatments (duration and dose)
Associated consumptions (decrease in using psychoactive substances) | 6 months
  GP will assessed and characterized other medical products taken in association with the treatment studied.

CONTACTS AND LOCATIONS:
Overall Officials: Maryse LAPEYRE-MESTRE, MD, Principal Investigator — University Hospital of Toulouse
Locations (5):
- France (5):
  - Clermont-Ferrand Hospital, Clermont-Ferrand
  - Grenoble Lyon Hospital, Grenoble
  - Marseille Hospital, Marseille
  - Nancy Hospital, Nancy
  - Service de Pharmacologie Médicale et Clinique - Centre d'addictovigilance - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dupouy J, Rousseau V, Authier N, Di Patrizio P, Gentile G, Gibaja V, Laporte C, Letrilliart L, Maynie C, Micallef J, Mallaret M, Oustric S, Berard E, Lapeyre-Mestre M. Impact of urine drug screening on opioid agonist treatment maintenance with buprenorphine in primary care in France: A cluster-randomized trial. Therapie. 2025 Jul 25:S0040-5957(25)00105-2. doi: 10.1016/j.therap.2025.07.003. Online ahead of print. PMID 40841272
- [Derived] ESUB-MG Study Group. Study protocol of the ESUB-MG cluster randomized trial: a pragmatic trial assessing the implementation of urine drug screening in general practice for buprenorphine maintained patients. BMC Fam Pract. 2016 Mar 1;17:24. doi: 10.1186/s12875-016-0413-3. PMID 26931763